CLINICAL TRIAL: NCT04201522
Title: The Effect of Respiratory Training With Normocapnic Hyperpnea on Exercise Tolerance in COPD
Brief Title: The Effect of Respiratory Training on Exercise Tolerance in COPD
Acronym: ERTET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Oueslati, Ferid, PhD (Unknown); Saey, Didier, M.D. (Individual)
Responsible Party: Principal Investigator, Francois Maltlais, Professor, MD, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CER 21411
Record Dates: First submitted 2019-11-26; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Respiratory training; COPD; Muscle oxygenation; Muscle fatigue; Oxygen kinetic; Exercise tolerance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: The study is a randomized, controlled, parallel-group trial.
Who Masked: Participant
Masking Description: Patients will be randomized to training group or sham group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training intervention (Active Comparator): The effect of 6-weeks of respiratory training with normocapnic hyperpnoea on exercise tolerance
  Interventions: Other: Normocapnic hyperpnoea intervention
- Sham intervention (Sham Comparator): The effect of 6-weeks of respiratory training with normocapnic hyperpnoea on exercise tolerance in the training group compared to the sham group.
  Interventions: Other: Sham intervention

INTERVENTIONS:
Other: Normocapnic hyperpnoea intervention — Patients will perform for 6-weeks, 15 min twice daily, 5 days a week at 60% of the peak of minute ventilation, at home by means of a respiratory device (SpiroTiger, Idiag, Fehraltorf, CH).
  Arms: Training intervention
Other: Sham intervention — Patients will perform for 6-weeks, 15 min twice daily, 5 days a week at rest's minute ventilation, at home by means of a respiratory device (SpiroTiger, Idiag, Fehraltorf, CH).
  Arms: Sham intervention

SUMMARY:
Exercise intolerance is one of the key disabling factors in patients with chronic obstructive pulmonary disease (COPD). Although multifactorial, exercise intolerance involves physiological interactions between respiratory and locomotor muscles that may contribute to further reducing exercise tolerance in COPD. The respiratory muscle work during exercise is closely related to breathing and could induce respiratory muscle fatigue in patients with COPD.

Respiratory muscle training is an intervention strategy that is sometimes proposed for some patients with COPD, especially whose with inspiratory muscle weakness. It was reported that inspiratory muscle training improves inspiratory muscle endurance and strength, dyspnea and exercise tolerance. There are two types of inspiratory muscle training, inspiratory muscle training against a resistive loading and normocapnic hyperpnoea. The advantage of normocapnic hyperpnoea compared to resistive training is the possibility to simulate the exercise ventilation level while maintaining stable the partial pressure of arterial carbon dioxide and end-tidal pressure of carbon dioxide and to solicit the inspiratory and expiratory muscles together, which could increase respiratory muscle tolerance and avoid their fatigue during whole-body exercise.

Therefore, the aim of this project is to study the effect of normocapnic hyperpnoea training on exercise tolerance in patients with COPD.

We hypothesize that greater improvement in cycling exercise tolerance will be observed following 6-weeks normocapnic hyperpnoea training compared to a sham intervention in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years;
* Chronic airflow obstruction : FEV1/FVC < 0.7, FEV1 of 30 to 80% predicted, after bronchodilation;

Exclusion Criteria:

* Inability to perform a cycling exercise;
* Diagnosed of one of more comorbidities that may limit exercise tolerance : cardiovascular, metabolic, endocrine, gastrointestinal, renal, neurological or rheumatologically disease;
* Recent COPD exacerbation (< 3 months);
* Recent cancer;
* A daily dose of Prednisone > 10 mg;
* Hypoxemia at rest or during exercise: PaO2 < 60 mmHg or SpO2 ≤ 88%;
* Body mass index > 30 kg/m²;
* Pregnancy;
* Skinfold at intercostal or vastus lateralis muscle > 1.5 cm.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-14 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Change in exercise tolerance (time [seconds]) | Baseline (week 0), 7 weeks
  Constant workrate cycling exercise time at 75% of power peak.

SECONDARY OUTCOMES:
Minute ventilation responses (flow [L/min]) | Baseline (week 0), 7 weeks
  Minute ventilation during the constant workrate cycling exercise will be determined using a portable gas analysis system.
Change in respiratory muscle strength (pressure [cm H2O]) | Baseline (week 0), 7 weeks
  Maximal inspiratory and expiratory pressures will be assessed with a portable manometer before and at end the constant workrate cycling exercise.
Change in muscle oxygenation (from baseline [%]) | Baseline (week 0), 7 weeks
  Deoxyhemoglobin/myoglobin concentrations measured by near-infrared spectroscopy of intercostal and vastus lateralis muscle during the constant workrate cycling exercise
Change in cardiac output (flow [L/min]) | Baseline (week 0), 7 weeks
  Arterial blood pressures and cardiac output will be non-invasively measured by a finger photoplethysmography device during the constant workrate cycling exercise
Isometric muscle strength (force [Kg]) | Baseline (week 0), 7 weeks
  Maximum voluntary isometric contraction with twitch tension induced by supramaximal magnetic stimulation of the femoral nerve will be realized before and 15 minutes after the constant workrate cycling exercise.

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec (IUCPQ)
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No